CLINICAL TRIAL: NCT00355966
Title: Comparison of Misorostol & PGE2 Gel for Immediate Induction of Labour for Premature Ropture of Membranes at Term
Brief Title: Comparison of Misoprostol and PGE2 Gel for Induction of Labour in Women With Premature Rupture of Membranes at Term
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nilratan Sircar Medical College (Other Government)
Responsible Party: Chairperson of Ethical Committee & Principal, Nilratan Sircar Medical College , Kolkata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Chaudhuri
Record Dates: First submitted 2006-07-18; First posted 2006-07-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2008-11

CONDITIONS: Premature Rupture of Membranes at Term
Keywords: Premature rupture of membranes; Induction of labour with Misoprostol; Induction of labour with PGE2 gel
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): In group A, immediate induction of labour will be done by intravaginal misoprostol 25 microgram 4 hourly , a maximum of 5 doses .
  Interventions: Drug: Misoprostol
- B (Active Comparator): In Group B immediate induction of labour will be done by application of vaginal PGE2 gel 0.5 gm at an interval of 6 hours , a maximum of 2 doses.
  Interventions: Drug: PGE2 gel

INTERVENTIONS:
Drug: Misoprostol — In one group of women immediate induction of labour will be done by intravaginal misoprostol 25 microgram 4 hourly , a maximum of 5 doses .
  Arms: A
Drug: PGE2 gel — In other group immediate induction of labour will be done by intravaginal application of PGE2 gel 0.5 mg at an interval of 6 hours , a maximum of 2 doses.
  Arms: B

SUMMARY:
Induction of labour with vaginal misoprostol, in women with premature rupture of membranes at term, results in significant shortening of induction to delivery time in comparison to vaginal PGE2 gel induction.

ELIGIBILITY:
Inclusion Criteria:

* Premature rupture of membranes at 37 or more weeks
* Single live fetus in cephalic presentation

Exclusion Criteria:

* Women in labour
* Women with contraindication of induction of labour
* Women with previous caesarean section or uterine surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Admission to delivery time | 48 hours

SECONDARY OUTCOMES:
Caesarean Section rate | 48 hours
Neonatal morbidity | Till discharge
Maternal morbidity | Till discharge

CONTACTS AND LOCATIONS:
Overall Officials: Snehamay Chaudhuri, MBBS,MD,DNB, Principal Investigator — NRS Medical College , Kolkata, India
Locations (1):
- NRS Medicl College,138 AJC Bose Road, Kolkata, West Bengal, India

REFERENCES:
- See also: Chaudhuri S, Mitra SN, Biswas PK, Bhattcharyya S.Pramature rupture of membranes at term: Immediate induction with PGE2 gel compared with delayed induction with oxytocin,Ind J Obstet Gynecol Vol56,no 3; 2006,224-229 — http://medind.nic.in/jaq/t06/i3/jaqt06i3p224.pdf